CLINICAL TRIAL: NCT02102373
Title: Clear Liquid vs Low-fiber Diet in Bowel Cleansing for Colonoscopy in Children: a Randomized Trial
Brief Title: Evaluation of Two Different Diet Regimen Prior to Colonoscopy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Aleksandra Banaszkiewicz, MD PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mytyk2014
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Children Prior to Colonoscopy
Keywords: colonoscopy, pediatric, preparation, diet

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- low-fiber diet (Active Comparator): Patients received low-fiber diet for 24 hours before colonoscopy
  Interventions: Device: polyethylene glycol 3350
- clear liquid diet (Active Comparator): Patients received clear liquid diet for 24 hours before colonoscopy
  Interventions: Device: polyethylene glycol 3350

INTERVENTIONS:
Device: polyethylene glycol 3350 — Patients received a polyethylene glycol 3350 solution starting at afternoon the day before the colonoscopy at a dose of 1000 ml/15 kg (maximum 4 L). The patients were instructed to drink all solution in about 4-6 hours.
  Other Names: Forlax

SUMMARY:
Colonoscopy is a routinely performed procedure in children and adolescents. Proper visualization of the intestinal mucosa is highly dependent on the quality of the bowel preparation. European Society of Gastrointestinal Endoscopy (ESGE) emphasizes that the timing of bowel preparation is the key factor and recommends that the delay between the last dose of bowel preparation and colonoscopy should be minimized. Timing of bowel preparation prior to colonoscopy has not been studied in children population, yet. The diet regimen before colonoscopy is likely less important than the timing of bowel preparation, however may influence the well-being of children.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years
* Elective colonoscopy

Exclusion Criteria:

* Chronic renal, liver, or heart failure
* Acute surgical abdominal conditions (e.g., acute obstruction or perforation)
* Acute surgical abdominal conditions (e.g., acute obstruction or perforation)
* Any prior gastrointestinal surgery

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Bowel preparation of the whole colon | in 15 minutes after colonoscopy
  Boston bowel preparation score for the whole colon assessed by the endoscopist in 15 minutes after the procedure

SECONDARY OUTCOMES:
Bowel preparation for colon sections | in 15 minutes after colonoscopy
  Boston bowel preparation score for:
  * the right side of the colon
  * the transverse section of the colon
  * the left side of the colon assessed by the endoscopist in 15 minutes after the colonoscopy
Duration of PEG taking | in 15 minutes after colonoscopy
Time between the last dose of PEG and colonoscopy | in 15 minutes after colonoscopy
Acceptability | in the first 6 hours after colonoscopy
  Patient's satisfaction of bowel preparation measured by 10-point visual-analogue scale (VAS)
Tolerability | in the first 6 hours after colonoscopy
  Tolerability assessment was based on the recording of occurrence and severity of GI symptoms such as nausea, bloating, abdominal, pain/cramps and anal discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Gastroenterology and Nutrition, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mytyk A, Lazowska-Przeorek I, Karolewska-Bochenek K, Kakol D, Banasiuk M, Walkowiak J, Albrecht P, Banaszkiewicz A. Clear Liquid Versus Low-fibre Diet in Bowel Cleansing for Colonoscopy in Children: A Randomized Trial. J Pediatr Gastroenterol Nutr. 2018 May;66(5):720-724. doi: 10.1097/MPG.0000000000001832. PMID 29112090
- See also: Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline — http://www.esge.com/assets/downloads/pdfs/guidelines/2013_bowel_preparation_for_colonoscopy.pdf